CLINICAL TRIAL: NCT04376255
Title: Augmented Reality Medical Simulation: A Multi-Collaborative Study of Acceptance and Usability
Brief Title: Augmented Reality Medical Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 55657
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Educational Problems
Keywords: Augmented Reality; Simulation; Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mixed Reality Simulation (Experimental): Participants in the experimental arm will be introduced to workplace training modules through an Augmented Reality (AR) headset.
  Interventions: Other: Augmented Reality (AR)

INTERVENTIONS:
Other: Augmented Reality (AR) — AR headset - a device that the participants will wear over their head and eyes and will add holographic elements to a live view of workplace training scenario

SUMMARY:
In order to improve the quality of care we provide to patients, medical trainees need to experience low incident, high mortality events in a safe learning environment. There is a selection bias for predisposing characteristics of health care providers, as most people who have pursued a career in medicine are motivated to learn how to manage medical emergencies. Resources have been traditionally enabled with conventional simulation centers or mobile simulation units. However, these are costly and difficult to access. The purpose of this study is to evaluate a mixed reality alternative to conventional simulation. The need for this is inherent in becoming a medical provider and use of these resources will improve health practices and health services.

ELIGIBILITY:
Inclusion Criteria:

* Trainees or personnel working and/or volunteering at Lucile Packard Children's Hospital Stanford / Stanford Health Care facilities
* 18 years and older

Exclusion Criteria:

* Have a history of severe motion sickness
* Currently have nausea
* History of seizures
* Are clinically unstable
* Currently using corrective glasses (not compatible with AR headset)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Qualitative Interview Assessment of Remote Simulations | Post-Simulation, Approximate time duration (3-5 minutes)
  Primary Aim: The primary aim is to study the acceptance of AR simulation among anesthesia residents using the Technology Acceptance Model (TAM)

SECONDARY OUTCOMES:
System Usability Scale (SUS) Questionnaire | Post-Simulation, Approximate time duration (3-5 minutes)
  The first secondary aim is to evaluate AR simulation usability via the System Usability Scale (SUS) and ISO 9241-400 Assessment of human-ergonomic factors.
Ergonomic Survey | Post-Simulation, Approximate time duration (3-5 minutes)
  : The final secondary aim will evaluate the ergonomics of the headset via the ISO 9241-400 Assessment of human-ergonomic factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States